CLINICAL TRIAL: NCT03680001
Title: Students Education Training in Emotional Connection
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G Welch, Associate Professor of Psychiatry in Pediatrics and Pathology & Cell Biology, Columbia University
Other Study IDs: AAAS0330
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Child Development; Premature Birth
Keywords: emotional connection; Martha G. Welch; nursing education
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Training in Rating Emotional Connection — Didactic education (video-supported educational module) on emotional connectivity will be offered to the subjects. Subjects will conference with PI to review ratings on modules.

SUMMARY:
The purpose of this study is to assess the effectiveness of different educational modules in training graduate students from Columbia University Irving Medical Center campus and from the Columbia School of Social Work to assess the emotional connection of mother/child dyads with accuracy.

The investigators hypothesize that after completing the educational module involving recorded dyad interactions, subjects will achieve coding reliability with the PI.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test educational modules designed to instruct students how to assess the quality and strength of mother-child relationships. The approach will use constructs of Emotional Connection that were used in development of an investigational observation-based screening instrument, the Welch Emotional Connection Screen (WECS). The WECS allows healthcare providers to rate the emotional connection of a mother-child relationship in just a few minutes of observed face-to face interaction, and shows preliminary predictive properties when performed in the first year of life.

Administration of the WECS involves watching recorded interactions of a child sitting face-to-face on the mother's lap, and scoring the interaction on sliding scales per 4 domains. During the WECS development, the Nurture Science Program of Columbia University Irving Medical Center created and coded hours of parent-child interaction videos. These videos will be used to assess and train the students (subjects) on rating mother/child dyads around emotional connection. Subjects will rate the quality of mother-child relationships in video training sets after completing one of two educational modules: A) a lecture-style webinar describing evidence base and instructions on how to score the WECS B) a guide written in Clear Explicit Translatable Language (CETL). Training set results of students in these groups will be compared to results of students who received no prior training. Training set results will be analyzed for the reliability statistic between student scores and key scores established by writer of the scale and PI. Subjects will then spend 3 months without further training in emotional connection or practice coding WECS. Subjects will then rate the quality of mother-child relationships for videos of dyads they hadn't previously seen. The main outcome of this study is the comparison of reliability statistics and maintenance between students who completed different educational modules.

ELIGIBILITY:
Inclusion Criteria:

* graduate students from the Columbia University Irving Medical Center campus and from the Columbia School of Social Work

Exclusion Criteria:

* refusal to participate

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Graduate students from the Columbia University Irving Medical Center campus and from the Columbia School of Social Work
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Intra-Class Correlations of Students' Welch Emotional Connection Screen (WECS) Scores | 2018 - 2019
  The Welch Emotional Connection Scale (WECS) is an investigational developmental screening tool, developed to rate the quality of the emotional connection that formed between mother and child. The scale is administered in 2-3 minutes by observing a mother and child interact, and requires the rater to critically assess 4 sub-domains of emotional connection.
  The WECS is scored on intervals of 0.25, with a minimum of 1 (little or no connection) and maximum of 3 (high connection). High connection is considered optimal for child development, and low connection is considered a risk in child development.
  Separately from these scores, the final portion of the screen determines, "Is the dyad emotionally connected?" and is scored with "No" or "Yes." Observing these scores could help determine if the educational module is successful in training students to assess the emotional connection.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Welch MG, Firestein MR, Austin J, Hane AA, Stark RI, Hofer MA, Garland M, Glickstein SB, Brunelli SA, Ludwig RJ, Myers MM. Family Nurture Intervention in the Neonatal Intensive Care Unit improves social-relatedness, attention, and neurodevelopment of preterm infants at 18 months in a randomized controlled trial. J Child Psychol Psychiatry. 2015 Nov;56(11):1202-11. doi: 10.1111/jcpp.12405. Epub 2015 Mar 11. PMID 25763525
- [Background] Hane AA, LaCoursiere JN, Mitsuyama M, Wieman S, Ludwig RJ, Kwon KY, V Browne J, Austin J, M Myers M, Welch MG. The Welch Emotional Connection Screen: validation of a brief mother-infant relational health screen. Acta Paediatr. 2019 Apr;108(4):615-625. doi: 10.1111/apa.14483. Epub 2018 Aug 13. PMID 29959878